CLINICAL TRIAL: NCT03695809
Title: Far Eastern Memorial Hospital
Brief Title: The Association of G9a Protein and Clinical Outcome of Patients With Vulvar Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 107008-F
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Vulvar Cancer, G9a Protein
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: G9a protein — To assess G9a protein expression on vulvar cancer

SUMMARY:
To assess the G9a expression in vulvar cancer

DETAILED DESCRIPTION:
Vulvar cancer can be treated with surgery, radiotherapy or chemoradiotherapy. Recurrence of vulvar cancer generally can be detected by imaging study. Currently, there is a paucity of sensitive marker to detect the recurrence of vulvar cancer. G9a is a recently identified protein with histone lysine methyltransferase activity. The role of histone methyltransferases in promoting tumorigenesis and progression of human cancers has been noted in some cancers, such as ovarian cancer, endometrial cancer and cervical cancer. The role of G9a protein in vulvar cancer remains obscure.

All female patients with vulvar cancer or vulvar intraepithelial neoplasm II /III who underwent surgery at Far Eastern Memorial Hospital from January 2003 will be included. All patients' clinical characteristerics including age, stage, pathologic finding, and follow-up data will be recorded from chart review.

The archived specimens will be used for immunohistochemical staining of G9a protein. Tumor size, local invasion, lymph node metastasis, and final disease stage will be determined. Correlation will be performed between G9a and clinical outcome of vulvar cancer.

ELIGIBILITY:
Inclusion Criteria:

* All female patients with vulvar cancer or vulvar intraepithelial neoplasm II /III who underwent surgery at Far Eastern Memorial Hospital from January 2003 were included.

Exclusion Criteria:

* N/A

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients' clinical characteristerics including age, stage, pathologic finding, and follow-up data were recorded from charts.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-04-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical outcome of vulvar cancer and G9a | 5 years
  The association of G9a protein and clinical outcome (such as overall survival and progression-free survival) of patients with vulvar cancer

SECONDARY OUTCOMES:
Correlation between histopathologic features of vulvar cancer and G9a | 1 year
  Correlation between histopathologic features (such as tumor grade, lymphovascular space invasion, lymph node metastasis and tumor size) of vulvar cancer and G9a

OTHER OUTCOMES:
Correlation between histopathologic features of vulvar intraepithelial neoplasm and G9a | 1 year
  Correlation between histopathologic features of vulvar intraepithelial neoplasm and G9a

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan